CLINICAL TRIAL: NCT00964678
Title: Pilot Study of the Safety and Efficacy of Carvedilol in Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM12120
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- carvedilol (Experimental): Carvedilol is titrated from a dose of 3.125mg twice daily to a maximal dose of 25mg twice daily over 24 weeks. Patients are evaluated to their response with 6 minute walk testing, echocardiography, and cardiac MRI
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Carvedilol — twice daily oral treatment in escalating dose
  Other Names: Coreg

SUMMARY:
The purpose of this study is to determine whether carvedilol treatment of patients with pulmonary arterial hypertension and associated right heart failure is safe and results in an improved function of the right heart.

DETAILED DESCRIPTION:
Patients with pulmonary arterial hypertension (PAH) will be treated with carvedilol for 24 weeks. During this time, carvedilol will be titrated from an initial dose of 3.125mg BID to a maximal dose of 25mg BID. At the start and end of the study, we will obtain cardiac MRI, 6 minute walk distance, brain natriuretic peptide (serum), echocardiogram, and functional class assessment. Our primary outcome is a change in right ventricular ejection fraction with cardiac MRI.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic, familial or associated PAH, WHO group 1
* NYHA class II or III
* clinically stable with optimized PAH treatment for at least 3 months
* no or minimal evidence of fluid overload or volume depletion, with or without diuretic treatment
* age > 18 years
* mean pulmonary artery pressure (mPAP) > 25 mmHg
* 6 minute walk distance (6MWD) over 100m

Exclusion Criteria:

* Structural heart disease unrelated to PAH
* Recent (<3 months) treatment with an intravenous positive inotropic agent
* current use of β-blockers
* history of reactive airways disease
* history of adverse reaction to β-blockers
* heart block on ECG or resting heart rate < 60 bpm
* cardiac index < 1.8 l/min/m2
* systemic hypotension (systolic pressure < 90 mmHg)
* pulmonary capillary wedge pressure > 15 mmHg
* inability to give informed consent
* contraindications to CT and/or PET scanning
* coagulopathy (INR>1.5 or platelet count<50000/mm3)
* severe renal insufficiency (creatinine clearance <30 ml/min/m2)
* malignancy or any co-morbidity limiting survival or conditions predicting inability to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C Grinnan, M.D, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared

REFERENCES:
- [Derived] Grinnan D, Bogaard HJ, Grizzard J, Van Tassell B, Abbate A, DeWilde C, Priday A, Voelkel NF. Treatment of group I pulmonary arterial hypertension with carvedilol is safe. Am J Respir Crit Care Med. 2014 Jun 15;189(12):1562-4. doi: 10.1164/rccm.201311-2025LE. No abstract available. PMID 24930531

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carvedilol
Started | 10
Completed | 6
Not Completed | 4
Not completed — Physician Decision | 4

BASELINE CHARACTERISTICS:
Population: Patients had pulmonary arterial hypertension, on pulmonary vasodilator therapy at baseline
Arm/Group | Carvedilol
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 60.6 [49 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 6
Right ventricular ejection fraction of blood [Mean (Full Range); unit: % of ejected ventricular vol of blood] | 38 [19 to 56]
Six minute walk distance [Mean (Full Range); unit: meters] | 321 [292 to 559]

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Right Ventricular Ejection Fraction
Description: Change in right ventricular ejection fraction is measured by cardiac magnetic resonance imaging, using the method of disks with the reading radiologist being blinded to before and after images. Cardiac magnetic resonance imaging was done at baseline and 6 months only
Time Frame: baseline, 6 months
Population: Patients with right heart catheterization confirmed pulmonary arterial hypertension, already on pulmonary vasodilator therapy
Measure: Mean (95% Confidence Interval); unit: % RVEF
Arm/Group | Carvedilol
Number analyzed (Participants) | 6
% RVEF | 10.4 [3.6 to 16]
Statistical Analysis 1: Comparison: Carvedilol; Test type: Superiority; p = 0.028, ANOVA — The threshold for statistical significance was p=0.05

2. Secondary Outcome: Change in Right Ventricular End Systolic Volume
Description: right ventricular end systolic volume determined by MRI
Time Frame: baseline and 6 months
Measure: Number; unit: mL
Arm/Group | Carvedilol
Number analyzed (Participants) | 6
mL
  Participant 1 | 3
  Participant 2 | 14
  Participant 3 | 56
  Participant 4 | 11
  Participant 5 | 27
  Participant 6 | 25
Statistical Analysis 1: Comparison: Carvedilol; Test type: Superiority; p = 0.028, ANOVA — The threshold for statistical significance was p=0.05

3. Secondary Outcome: Change in 6 Minute Walk Distance
Time Frame: baseline and 6 months
Population: The patient who was excluded from analysis developed an orthopedic injury during the study and was unable to complete the walking test at conclusion of the study
Measure: Number; unit: feet
Arm/Group | Carvedilol
Number analyzed (Participants) | 5
feet
  Participant 1 | 45
  Participant 2 | 160
  Participant 3 | 35
  Participant 5 | 5
  Participant 6 | 96
Statistical Analysis 1: Comparison: Carvedilol; Test type: Superiority; p > 0.05, ANOVA — The threshold for statistical significance was p=0.05

4. Secondary Outcome: Change in Tricuspid Annular Plane Systolic Excursion
Description: Higher values indicate a better outcome.
Time Frame: baseline and 6 months
Population: The patient excluded from the analysis was unable to be present for the final echo-cardiogram due to lack of transportation and distance from the hospital. Multiple attempts to schedule the study test were made through phone and email.
Measure: Number; unit: centimeters
Arm/Group | Carvedilol
Number analyzed (Participants) | 5
centimeters
  Participant 1 | 0.4
  Participant 2 | -0.08
  Participant 4 | -0.12
  Participant 5 | 0.45
  Participant 6 | 0.08
Statistical Analysis 1: Comparison: Carvedilol; Test type: Superiority; p > 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Carvedilol
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carvedilol (N=6)
fatigue (Metabolism and nutrition disorders) | 1 (1) — mild, resolved with dose reduction and slow rate of titration
hypotension (Cardiac disorders) | 1 (1) — asymptomatic. Mild, resolved with dose reduction

LIMITATIONS AND CAVEATS:
Small number of patients enrolled. This study is hypothesis generating and was meant to lead to larger studies of carvedilol in pulmonary hypertension

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No